CLINICAL TRIAL: NCT02011399
Title: EEG-based Brain Computer Interface and Mu Rhythm for Computer Access
Brief Title: Brain Computer Interfaces (Mu Rhythm Learning)
Status: Terminated | Type: Observational
Why Stopped: Training procedure was not effective.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Assistant Professor, University of Michigan
Other Study IDs: I0001
Record Dates: First submitted 2011-04-15; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Mobility Impairments
Keywords: brain; computer; interfaces; mobility impairments
MeSH Terms: interventions — Brain-Computer Interfaces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Brain Computer Interface for Mu Rhythm — Device: Brain Computer Interface Subjects will wear an EEG (electrode) cap for 1-4 hours (1-2 hours typical) per session and use the brain-computer interface to operate a computer. Subjects will be asked to participate in 4-20 sessions.
  Arms: Brain Computer Interface Keyboard
  Other Names: The electrode cap used is made by Electro-cap International.

SUMMARY:
Sensorimotor (also know as mu) rhythm based brain-computer interfaces (BCIs) are a tool for controlling electronic devices using only brain signals.

The Mu rhythm is a naturally occuring wave produced by the brain. This research project will determine how to best train subjects to use the Mu rhythm for computer control.

DETAILED DESCRIPTION:
As a method of BCI control, Mu rhythms are difficult to learn and involve extensive training. The investigators want to keep users motivated and determine the best way to provide effective training. Healthy users will be trained to control a computer by wearing an electrode cap that is connected to a computer. They will have their levels of motivation and interest measured while learning to use the Mu rhythm. Two different types of learning programs will be used to determine which is most effective for Mu rhythm training. This method will be used for device control by people with severe physical impairments, who may be able to communicate or carry out other desired tasks using a BCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Able to read text on a computer screen
* Able to understand and remember instructions concerning participation

Exclusion Criteria:

* Unable give informed consent.
* Unable to understand and follow instructions.
* Have abnormal tone or uncontrolled movements in the head-and-neck that would interfere with EEG recordings.
* Known to have photosensitive epilepsy.
* Open head lesions or sores

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Mu Rhythm Learning | 20 sessions
  The primary outcome measure is determining the best learning methods by which subjects can learn to use the Mu rhythm to hit targets on a computer screen.

CONTACTS AND LOCATIONS:
Overall Officials: Jane E. Huggins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States